CLINICAL TRIAL: NCT07324720
Title: Strategic Comparison Of Ischemia-based Versus Plaque Burden and vulnErability-based Revascularization in High-Risk Coronary Artery Disease Patients
Acronym: SCOPE-HR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bon-Kwon Koo (Other)
Collaborators: Biotronik Korea Co., Ltd (Industry); COBEMD (Unknown)
Responsible Party: Sponsor-Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2508-177-1673
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plaque burden and vulnerability-based revascularization (Experimental): Percutaneous coronary intervention using drug-eluting stent(s) will be performed by IVUS or OCT-guided strategy.
  Interventions: Procedure: Plaque burden and vulnerability-based revascularization
- Ischemia-based revascularization (Active Comparator): Percutaneous coronary intervention using drug-eluting stent(s) will be performed by FFR, iFR, or angiography-derived FFR-guided strategy.
  Interventions: Procedure: Ischemia-based revascularization

INTERVENTIONS:
Procedure: Plaque burden and vulnerability-based revascularization — For target lesions located in vessels with a reference diameter ≥2.5 mm, quantitative and qualitative plaque assessment will be performed using intravascular imaging. The criteria for revascularization are as follows:
  1. When using IVUS:
     Revascularization will be considered for lesions with a minimum lumen area (MLA) < 4 mm² if any of the following findings are present:
     * Plaque burden > 70%
       * Plaque rupture ③ Thrombosis ④ Posterior attenuation without high-intensity echo reflectors (involving > 180° of the vessel circumference) ⑤ maxLCBI₄mm > 315 on near-infrared spectroscopy (NIRS)
  2. When using OCT:
  Revascularization will be considered for lesions with a minimum lumen area (MLA) < 3.5 mm² if any of the following findings are present:
  * Area stenosis ≥ 75%
    * Plaque rupture
      * Presence of a thin fibrous cap < 65 μm ④ Lipid arc > 180° ⑤ Macrophage infiltration
  During revascularization, the operator should ensure optimal treatment of the target vessel and lesion, using intravascular
  Arms: Plaque burden and vulnerability-based revascularization
Procedure: Ischemia-based revascularization — For target lesions located in vessels with a reference diameter ≥2.5 mm, the presence or absence of myocardial ischemia will be evaluated using FFR, iFR, or angiography-derived FFR. The criteria for revascularization are as follows:
  1. Lesions with ≥50% diameter stenosis by visual estimation and FFR ≤ 0.80
  2. Lesions with ≥50% diameter stenosis by visual estimation and iFR < 0.89
  3. Lesions with ≥50% diameter stenosis by visual estimation and angiography-derived FFR ≤ 0.80
  During revascularization, the operator should ensure optimal treatment of the target vessel and target lesion, utilizing intravascular imaging modalities such as IVUS or OCT. The criteria for optimal revascularization are as follows, and operators are strongly encouraged to achieve them:
  1. For all treated vessels, achieve post-PCI FFR > 0.86, with a minimum threshold of post-PCI FFR > 0.80, to ensure functionally complete revascularization.
  2. Achieve post-PCI ΔFFR ([FFR at the stent distal edge] - [FFR at the s
  Arms: Ischemia-based revascularization

SUMMARY:
1. Study Purpose This study aims to compare clinical outcomes between two revascularization strategies in patients with high-risk coronary artery disease and 50-90% angiographic stenosis: a plaque burden and vulnerability-based revascularization strategy guided by intravascular imaging versus an ischemia-based revascularization strategy guided by physiologic assessment.
2. Background Percutaneous coronary intervention (PCI), in conjunction with optimal medical therapy, is one of the main therapeutic strategies for improving outcomes in patients with CAD. To enhance the results of PCI, various diagnostic and adjunctive techniques have been developed-most notably, invasive physiologic assessment and intravascular imaging (IVI). Invasive physiologic indices such as fractional flow reserve (FFR) and instantaneous wave-free ratio (iFR) are recognized as the most accurate methods to determine vessel-level myocardial ischemia, and current guidelines recommend PCI based on these physiological measurements. Recently, angiography-derived FFR has also been developed, allowing ischemia assessment without pressure wire measurement, and has been endorsed as a useful tool for guiding PCI decisions. Intravascular imaging, on the other hand, provides detailed anatomical insights into atherosclerotic plaque morphology and plays a critical role in achieving procedural optimization. Current guidelines recommend the use of IVI, particularly in the treatment of complex lesions. While most previous IVI studies have focused on procedural optimization, more recent investigations have begun to explore the use of IVI for PCI decision-making itself. Emerging data suggest that revascularization decisions based on quantitative and qualitative plaque assessment using IVI are non-inferior to those based on invasive physiologic testing. Moreover, IVI enables the identification of vulnerable plaques, and studies indicate that intervening on such lesions may improve outcomes.

   At present, a physiology-guided decision-making strategy combined with IVI-guided optimization is considered the best evidence-based approach according to guidelines. However, recent data showing the potential advantages of IVI-guided decision-making and IVI-guided optimization-particularly in high-risk, complex patients and in those with vulnerable plaque morphology-suggest that IVI-based strategies may offer greater clinical benefit in such populations. Despite this, a comprehensive strategy that integrates both quantitative (plaque burden) and qualitative (vulnerability) aspects of plaque evaluation via IVI has yet to be clearly established. Therefore, this study seeks to propose IVI-based quantitative and qualitative criteria for high-risk CAD patients and to compare outcomes between a plaque burden and vulnerability-based revascularization strategy and the conventional ischemia-based revascularization strategy. For all patients undergoing PCI, IVI-guided optimization will be performed to ensure the highest possible procedural quality in both groups.
3. Study Procedures Patients undergoing coronary angiography for suspected or known CAD will be screened for eligibility. After providing a detailed explanation of the study, written informed consent will be obtained from those deemed appropriate for participation. Following coronary angiography, patients with significant coronary stenosis who meet all inclusion and no exclusion criteria will be enrolled in the study. Eligible participants will then be randomized in a 1:1 ratio to either the plaque burden and vulnerability-based revascularization group or the ischemia-based revascularization group. Stratified randomization will be performed according to participating center and presence or absence of acute coronary syndrome (ACS) to ensure balance between the groups.

ELIGIBILITY:
Inclusion Criteria:

① Patients aged 19 years or older

② Patients with moderate to severe coronary artery stenosis identified on coronary angiography:

A. Diameter stenosis of 50%-90% by visual estimation B. De novo lesions (newly developed lesions) C. Reference vessel diameter ≥ 2.5 mm by visual estimation

③ Patients with either clinically high-risk features for recurrent ischemic events or complex high-risk lesions identified on angiography:

A. Clinically high-risk features i. Medically treated diabetes mellitus ii. Chronic kidney disease (≥ Stage 3B, eGFR < 45 mL/min/1.73 m²) iii. Acute coronary syndrome (ACS) iv. Previous myocardial infarction (MI)

B. Complex high-risk lesions i. True bifurcation lesions ii. Calcified lesions (moderate to severe calcification on angiography) iii. Diffuse long lesions (≥ 30 mm in length) iv. Multivessel disease v. Multiple lesions (≥ 3 lesions)

④ Patients who can verbally demonstrate an understanding of the risks, benefits, and alternative treatments of invasive physiologic or imaging assessment and PCI

⑤ Patients who agree to the study protocol and clinical follow-up plan, voluntarily decide to participate, and provide written informed consent to participate in this clinical trial

Exclusion Criteria:

* Hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, prasugrel, ticagrelor, adenosine, or nicorandil

  * Hemodynamic instability requiring mechanical circulatory support (ECMO or IABP)

    * Moderate or severe stenosis of the left main coronary artery (diameter stenosis > 50%)

      * History of coronary artery bypass grafting (CABG)

        * Severe asthma or severe chronic obstructive pulmonary disease (COPD) ⑥ Active bleeding

          ⑦ Major gastrointestinal or genitourinary bleeding within the previous 3 months

          ⑧ Bleeding diathesis or known coagulopathy, including a history of heparin-induced thrombocytopenia (HIT)

          ⑨ Life expectancy < 2 years due to non-cardiovascular comorbidities

          ⑩ Inability to provide signed informed consent

          ⑪ Any condition deemed by the investigator to make the patient unsuitable for this clinical trial or likely to increase study-related risks

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1944 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2033-09-24 (Estimated); Study Completion 2033-09-24 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure | 2 years after last patient enrollment
  a composite of cardiovascular death, target vessel myocardial infarction and ischemia-driven target vessel revascularization

SECONDARY OUTCOMES:
Patient-oriented composite outcome | 2 years after last patient enrollment
  a composite of all cause of death, any myocardial infarction and any repeat revascularization
Target lesion failure | 2 years after last patient enrollment
  a composite of cardiovascular death, target vessel myocardial infarction and ischemia-driven target lesion revascularization
All cause death | 2 years after last patient enrollment
Cardiovascular death | 2 years after last patient enrollment
Any myocardial infarction | 2 years after last patient enrollment
Peri-procedural myocardial infarction | 3 days after procedure
Target vessel myocardial infarction | 2 years after last patient enrollment
Definite or probable stent thrombosis | 2 years after last patient enrollment
Ischemic or hemorrhagic stroke | 2 years after last patient enrollment
Any revascularization | 2 years after last patient enrollment
Ischemia-driven target vessel revascularization | 2 years after last patient enrollment
Ischemia-driven target lesion revascularization | 2 years after last patient enrollment
Number of stents used per patient or lesion | After procedure
Bleeding Academic Research Consortium [BARC] type 2,3, or 5 | 2 years after last patient enrollment

IPD SHARING:
Plan to Share IPD: No